CLINICAL TRIAL: NCT04881968
Title: Hopewell Hospitalist: A Video Game Intervention to Increase Advance Care Planning Conversations by Hospitalists With Older Adults
Brief Title: EFFECTIVENESS: Hopewell Hospitalist: A Video Game Intervention to Increase Advance Care Planning by Hospitalists
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The effectiveness trial was terminated early because the intervention proved to be ineffective in generating engagement from study participants. With such low engagement we were unable to test our intervention with our proposed outcome measures.
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Sound Physicians (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Amber Barnato, Susan J. and Richard M. Levy 1960 Distinguished Professor in Health Care Delivery, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00031186 - B; P01AG019783 (NIH)
Record Dates: First submitted 2021-05-06; First posted 2021-05-11 (Actual); Results first posted 2022-02-02 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Advance Care Planning
Keywords: advance care planning; physician performance; serious games; narrative engagement

STUDY DESIGN:
Intervention Model Description: We will email the Uniform Resource Locator (URL) to download the App with encouragement to play the game, including positive feedback from participants in the efficacy study. Receipt of the email will be our measure of intervention delivery. Each hospitalist 'crosses over' from control to intervention at a single time point.
Who Masked: Outcomes Assessor
Masking Description: A physician's treatment assignment will be masked during analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: Usual Care (No Intervention): The control arm occurs prior to receipt of the video game intervention and reflects usual care. Each hospitalist 'crosses over' from control to intervention at a single time point.
- Video Game Intervention (Experimental): Each hospitalist 'crosses over' from control to intervention at a single time point by receiving a link to the Hopewell Hospitalist game via email and logging in to play the video game.
  Interventions: Behavioral: Hopewell Hospitalist Video Game

INTERVENTIONS:
Behavioral: Hopewell Hospitalist Video Game — Hopewell Hospitalist is a customized theory-based adventure video game that uses narrative engagement to educate physician players on advance care planning to increase physicians' likelihood of engaging in and billing for ACP conversations.
  Arms: Video Game Intervention

SUMMARY:
Hopewell Hospitalist is a theory-based adventure video game designed to increase the likelihood that a physician will engage in an advance care planning (ACP) conversation with a patient over the age of 65. Drawing on the theory of narrative engagement, players assume the persona of a hospitalist physician and navigate a series of clinical encounters with seriously-ill patients over the age of 65. Players experience the consequences of having (or not having) ACP conversations in a timely fashion. The planned study is a crossover phase III trial testing the effectiveness of providing physicians with a link to a free version of Hopewell Hospitalist as a means for increasing ACP rates measured by ACP billing frequency.

ELIGIBILITY:
Hospitalist Inclusion Criteria:

* Employed by Sound
* Not previously included in the Efficacy Trial Arm of the study.

Hospitalist Exclusion Criteria:

* Not employed by Sound
* Does not provide informed consent
* Previously included in the Efficacy Trial Arm of the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1261 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amber Barnato, MD, MPH, MS, Principal Investigator — Dartmouth-Hitchcock Medical Center and Geisel School of Medicine�
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified participant data and supporting information with other researchers upon request to the PI.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon publication of the planned manuscripts. Data will be retained through February 2028.
Access Criteria: Data will require completion of a data use agreement with Dartmouth.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Individuals who received an invitation via an email from the Chief Experience Officer at Sound Physicians were considered enrolled. In this pre/post study design, each participant would be assigned to both the Control Arm, in which we would analyze ACP billing 90 days prior to the intervention, and the Video Game Intervention Arm, in which we would analyze ACP billing 90 days post intervention.
Groups:
- Entire Study Population: Each hospitalist in our study population 'crosses over' from control to intervention at a single time point by receiving a link to the Hopewell Hospitalist game via email and logging in to play the video game.
  Hopewell Hospitalist Video Game: Hopewell Hospitalist is a customized theory-based adventure video game that uses narrative engagement to educate physician players on advance care planning to increase physicians' likelihood of engaging in and billing for ACP conversations.
Period: Overall Study
Arm/Group | Entire Study Population
Started | 1261
Completed | 1261
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 1261
Age, Customized [Number; unit: participants] — We did not collect information regarding age from study participants. Population: We did not collect information regarding age from study participants.
Sex: Female, Male [Count of Participants; unit: Participants] — We did not collect information regarding sex from study participants. Population: We did not collect information regarding sex from study participants.
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — We did not collect information regarding race/ethnicity from study participants. Population: We did not collect information regarding race/ethnicity from study participants.
Region of Enrollment [Number; unit: participants]
  United States | 1261

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Billed Advance Care Planning
Description: Change in physician advance care planning billing for patients over the age of 65 in the three months before and after the roll-out of the video game intervention at their hospital. Advance care planning billing is defined as the presence/absence of ACP charges (Medicare billing codes 99497 or 99498) during a physician's patient's hospitalization.
Time Frame: 6 months (3 months pre and 3 months post intervention)
Population: We are reporting on all study participants in this section. No data was collected for the Primary Outcome: Incidence of Billed Advance Care Planning.
Groups:
- Pre/Post Arms Combined: This covers both pre and post arms proposed in our study.
Arm/Group | Pre/Post Arms Combined
Number analyzed (Participants) | 0

2. Primary Outcome: Merit-based Incentive Payment System Advance Care Planning Quality Score
Description: Change in the Merit-based Incentive Payment System (MIPS) self-report measure of advance care planning by enrolled hospitalists (MiPS-ACP quality score). The MiPS-ACP quality score is the percentage of patients aged 65 years and older who have an advance care plan or surrogate decision maker documented in the medical record or documentation in the medical record that an advance care plan was discussed but the patient did not wish or was not able to name a surrogate decision maker or provide an advance care plan. The quality score ranges from 0-100%, with higher scores indicating that a greater proportion of patients with an advance care plan documented in the medical record.
Time Frame: 6 months (3 months pre and 3 months post intervention)
Population: We are reporting on all study participants in this section. No data was collected for the Primary Outcome: Merit-based Incentive Payment System Advance Care Planning Quality Score.
Arm/Group | Pre/Post Arms Combined
Number analyzed (Participants) | 0

3. Secondary Outcome: Hospitalist-Managed Patient In-Hospital Mortality Rate
Description: In-hospital mortality rate for patients managed by enrolled hospitalists.
Time Frame: 6 months (3 months pre and 3 months post intervention)
Population: We are reporting on all study participants in this section. No data was collected for the Secondary Outcome: Hospitalist-Managed Patient In-Hospital Mortality Rate.
Arm/Group | Pre/Post Arms Combined
Number analyzed (Participants) | 0

4. Secondary Outcome: Hospitalist-Managed Patient 90-Day Mortality Rate
Description: 90-day mortality rate for patients managed by enrolled hospitalists.
Time Frame: 6 months (3 months pre and 3 months post intervention)
Population: We are reporting on all study participants in this section. No data was collected for the Secondary Outcome: Hospitalist-Managed Patient 90-Day Mortality Rate.
Arm/Group | Pre/Post Arms Combined
Number analyzed (Participants) | 0

5. Secondary Outcome: Sum of Resources Utilized by Hospitalist-Managed Patients
Description: Combined sum of resources utilized by patients managed by enrolled hospitalists during their index hospitalization (first hospitalization in the relevant period: control or intervention). It is a composite measure including: admission to ICU, receipt of life-sustaining treatment(s) including mechanical ventilation, placement of tracheostomy, insertion of gastric feeding tube, new onset dialysis. This measure ranges from 0 to 5, where higher scores indicate greater utilization of resources during the index hospitalization.
Time Frame: 6 months (3 months pre and 3 months post intervention)
Population: We are reporting on all study participants in this section. No data was collected for the Secondary Outcome: Sum of Resources Utilized by Hospitalist-Managed Patients.
Arm/Group | Pre/Post Arms Combined
Number analyzed (Participants) | 0

6. Secondary Outcome: Incidence of Hospitalist-Managed Patient Admission to ICU
Description: Incidence of admission to ICU for patients managed by enrolled hospitalists during their index hospitalization (first hospitalization in the relevant period: control or intervention).
Time Frame: 6 months (3 months pre and 3 months post intervention)
Population: We are reporting on all study participants in this section. No data was collected for the Secondary Outcome: Incidence of Hospitalist-Managed Patient Admission to ICU.
Arm/Group | Pre/Post Arms Combined
Number analyzed (Participants) | 0

7. Secondary Outcome: Incidence of Hospitalist-Managed Patient Mechanical Ventilation
Description: Incidence of mechanical ventilation of patients managed by enrolled hospitalists during their index hospitalization (first hospitalization in the relevant period: control or intervention).
Time Frame: 6 months (3 months pre and 3 months post intervention)
Population: We are reporting on all study participants in this section. No data was collected for the Secondary Outcome: Incidence of Hospitalist-Managed Patient Mechanical Ventilation.
Arm/Group | Pre/Post Arms Combined
Number analyzed (Participants) | 0

8. Secondary Outcome: Incidence of Hospitalist-Managed Patient Receipt of Life-Sustaining Treatment(s)
Description: Incidence of placement of tracheostomy, insertion of gastric feeding tube, new onset dialysis for patients managed by enrolled hospitalists during their index hospitalization (first hospitalization in the relevant period: control or intervention).
Time Frame: 6 months (3 months pre and 3 months post intervention)
Population: We are reporting on all study participants in this section. No data was collected for the Secondary Outcome: Incidence of Hospitalist-Managed Patient Receipt of Life-Sustaining Treatment(s).
Arm/Group | Pre/Post Arms Combined
Number analyzed (Participants) | 0

9. Secondary Outcome: Hospitalist-Managed Patient Length of Stay
Description: Total days between admission and discharge for patients managed by enrolled hospitalists.
Time Frame: 6 months (3 months pre and 3 months post intervention)
Population: We are reporting on all study participants in this section. No data was collected for the Secondary Outcome: Hospitalist-Managed Patient Length of Stay
Arm/Group | Pre/Post Arms Combined
Number analyzed (Participants) | 0

10. Secondary Outcome: Hospitalist-Managed Patient Disposition Status Type
Description: Type of status upon discharge of patients managed by enrolled hospitalists (e.g., discharged to home, to skilled nursing, to hospice, deceased, etc.).
Time Frame: 6 months (3 months pre and 3 months post intervention)
Population: We are reporting on all study participants in this section. No data was collected for the Secondary Outcome: Hospitalist-Managed Patient Disposition Status Type
Arm/Group | Pre/Post Arms Combined
Number analyzed (Participants) | 0

11. Secondary Outcome: Hospitalist-Managed Patient 90-Day Episode-Based Spending
Description: Amount of total Medicare payments between index admission and 90-days for patients managed by enrolled hospitalists.
Time Frame: 6 months (3 months pre and 3 months post intervention)
Population: We are reporting on all study participants in this section. No data was collected for the Secondary Outcome: Hospitalist-Managed Patient 90-Day Episode-Based Spending
Arm/Group | Pre/Post Arms Combined
Number analyzed (Participants) | 0

12. Other Pre Specified Outcome: Hopewell Hospitalist - Apple App Store and Google Analytics
Description: Number of unique downloads for the HH game will be provided by the Apple App store. Using Google Analytics we will be able to discern time spent playing the game for each individual hospitalist using their unique log-in passphrase.
Time Frame: 3 months
Population: We are reporting on all study participants in this section. No data was collected for the Secondary Outcome: Hopewell Hospitalist - Apple App Store and Google Analytics
Arm/Group | Pre/Post Arms Combined
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events information was not collected during this study. The intervention involved two emails sent to physicians at eligible Sound Hospitals containing a link to an educational video game.
Description: Total Number of Participants at Risk is zero (0) as mortality, serious and other [non-serious] adverse events were not collected or assessed as part of the study.
Groups:
- Entire Study Population: Adverse events information was not collected during this study.
Arm/Group | Entire Study Population
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/68/NCT04881968/Prot_SAP_000.pdf